CLINICAL TRIAL: NCT02600221
Title: A Non-interventional Study to Investigate the Current Situation of Asthma-COPD Overlap Syndrome in Patients Over Age 40 With Persistent Airflow Limitation in China
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00102
Record Dates: First submitted 2015-10-29; First posted 2015-11-09 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Asthma-COPD Overlap Syndrome
Keywords: ACOS
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the distributions of the patients with ACOS, asthma and COPD over age 40 with chronic airflow limitation in China.

DETAILED DESCRIPTION:
Sites must be tier 3 hospitals in China. Investigators will mainly be determined according to the following criteria:

* Respiratory physicians working in the respiratory department of tier 3 hospitals
* To include the expected number of patients in a maximum of 12 months, physicians should manage a reasonable number of asthma, COPD or ACOS over age 40 with persistent airflow limitation (post-BD FEV1/FVC<0.7).
* Physicians should have patients' spirometric data available in the patient's medical files (post-BD FEV1%pred and post-BD FEV1/FVC).

This NIS will collect the data (e.g. medical record, patient or physician-reported data) from about 2000 consecutive outpatients with persistent airflow limitation(post-BD FEV1/FVC<0.7) in about 20 sites in China for one year. Each site will recruit about 50-150 patients successively.

The data will be collected under routine clinical practice. The treatments or examinations will be determined by their treating physicians. The data are expected to reflect the actual situation about ACOS.

The study population will be about 2000 outpatients, men or women, over age 40, with a clinical diagnosis of asthma, COPD or ACOS with persistent airflow limitation（post-BD FEV1/FVC<0.7）in China from Q4,2015 to Q3,2016.

ELIGIBILITY:
Inclusion Criteria:

Outpatients, age ≥ 40 years Clinically diagnosed as asthma, COPD/chronic bronchitis/emphysema or ACOS at least 12 months With persistent airflow limitation (post-BD FEV1/FVC<0.7) Signed informed consent forms

Exclusion Criteria:

Have been involved in other clinical trial within 3 months Having other respiratory diseases which can influence airflow, such as lung cancer, tuberculosis, pneumonia, bronchiectasis, etc With acute exacerbation Inability to understand the study procedures or inability/reluctance to answer questionnaire judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be about 2000 outpatients, men or women, over age 40, with a clinical diagnosis of asthma, COPD or ACOS with persistent airflow limitation（post-BD FEV1/FVC<0.7）in China from Q4,2015 to Q3,2016.
Sampling Method: Non-Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
The proportion of ACOS among the patients over age 40 with persistent airflow limitation (post-BD FEV1/FVC<0.7) based on GINA and GOLD 2015 definition | one day

SECONDARY OUTCOMES:
- The proportions of COPD and asthma, respectively, among the patients over age 40 with persistent airflow limitation (post-BD FEV1/FVC<0.7) based on GINA and GOLD 2015 definition. | one day
- The distributions of the severity of airflow limitation according to GOLD lung function grading based on post-BD FEV1 in patients with ACOS, COPD or asthma. | one day
- The distribution of groups according to GOLD 2015 group definition (A,B,C,D) in patients with ACOS or COPD. | one day
- The distribution of medication by drug class in patients with ACOS, Asthma and COPD. | one day
- The proportions of previous diagnosis as asthma/COPD/chronic bronchitis/emphysema in the ACOS patients. | one day
The number of Acute exacerbations history in 12 months before the visit | one day
The severity of Acute exacerbations history in 12 months before the visit | one day
The days of hospitalization or emergency room visit of Acute exacerbations history in 12 months before the visit | one day
Severity of ACOS patients evaluated using CAT (mild, moderate, severe and very severe) in ACOS patients | one day
Severity of ACOS patients evaluated using ACQ-5 (complete control, good control and uncontrolled) in ACOS patients | one day
Severity of ACOS patients evaluated using mMRC (0, 1, 2, 3 and 4) in ACOS patients | one day

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kang, Doctor of Medicine, Principal Investigator — First Hospital of China Medical University
Locations (13):
- China (13):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Haikou, Hainan
  - Research Site, Zhengzhou, Henan
  - Research Site, Changsha, Hunan
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdou, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Kang J, Zheng J, Cai B, Wen F, Yao W, Zhang X, Chen Y, Wang G, Li W, Cao J. Current situation of asthma-COPD overlap in Chinese patients older than 40 years with airflow limitation: a multicenter, cross-sectional, non-interventional study. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620961699. doi: 10.1177/1753466620961699. PMID 33103591
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3996&filename=ACOS_CSR_synopsis.pdf